CLINICAL TRIAL: NCT01398748
Title: A Phase 1 Study of Intranasal Reduced Glutathione in Parkinson's Disease
Brief Title: Intranasal Glutathione in Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bastyr University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BU-H32B11; 5K01AT004404 (NIH)
Record Dates: First submitted 2011-07-19; First posted 2011-07-21 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Parkinson's Disease (PD)
Keywords: Parkinson's disease; Neuroprotection; Glutathione; Intranasal
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Intranasal GSH 100mg/ml (Active Comparator): Study participant will be provided with monthly supply of study medication and will be asked to intake 100mg/ml of intranasal glutathione (n=15) An amount of 1ml with a frequency 3x per days and duration of 12 weeks with a dosage of 2100mg
  Interventions: Drug: Intranasal glutathione - (in)GSH
- Intranasal glutathione 200mg/ml (Active Comparator): Study participant will be provided with monthly supply of study medication and will be asked to intake 200/ml of intranasal glutathione (n=15) An amount of 1ml with a frequency 3x per days and duration of 12 weeks with a dosage of 4200mg
  Interventions: Drug: Intranasal glutathione - (in)GSH
- Saline intranasal delivery (Placebo Comparator): Study participant will be provided with monthly supply of study medication and will be asked to intake Intranasal saline delivery (n=15) An amount of 1ml with a frequency 3x per day with a duration of 12 weeks
  Interventions: Drug: Saline Intranasal Delivery
- Watchful waiting (No Intervention): No intervention, watchful waiting only (n=4)

INTERVENTIONS:
Drug: Intranasal glutathione - (in)GSH — Intranasal glutathione-Tripeptide glutathione 100 mg/ml. 1 ml 3x per day TID X 12 weeks at 2100mg in 15 participants
  Arms: Intranasal GSH 100mg/ml
Drug: Intranasal glutathione - (in)GSH — Intranasal Glutathione-Tripeptide glutathione - 200mg/ml. 1 ml 3x per day TID X 12 weeks at 4200mg in 15 participants
  Arms: Intranasal glutathione 200mg/ml
Drug: Saline Intranasal Delivery — Saline administration 1ml 3x/day 12 weeks in 15 participants
  Arms: Saline intranasal delivery

SUMMARY:
Excessive free radical formation and depletion of the brain's primary antioxidant, glutathione, are established components of Parkinson's disease (PD) pathophysiology. While there is rationale for the therapeutic use of reduced glutathione (GSH) in PD, and even some preliminary evidence to suggest the use of GSH can lead to symptomatic improvement, obstacles surrounding currently employed delivery methods have hindered the clinical utility of this therapy. Intranasal GSH, (in)GSH, is a novel method of delivery for this popular CAM therapy in patients with PD, and bypasses the obstacles associated with other delivery methods. It has been used in clinical practice since 2005. The aim of this study is to evaluate safety, tolerability, and preliminary absorption data of (in)GSH in volunteers with PD in a Phase I single ascending dose escalation study.

DETAILED DESCRIPTION:
Individuals will be randomized to one of three treatment (100 mg GSH/ ml, 200 mg GSH/ ml, or placebo) arms in a double-blind fashion. All study medication will be administered 1 ml three times daily for three months, with a one-month wash out.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Parkinson's Disease made by neurologist within previous 10 years
2. Modified Hoehn and Yahr Stage <3
3. Age >20
4. Subjects must be able to attend study visits at screening, baseline, weeks 4, 8, 12, 16
5. Subjects must be able to demonstrate self-administration of study medication or have active caregiver who can administer daily.
6. Dose and frequency of all pharmaceutical medications must be stable for one month prior to enrollment.
7. Diet, exercise and supplementation must be kept constant throughout participation in study
8. Ability to read and speak English

Exclusion Criteria:

1. Dementia as evidenced by Montreal Cognitive Assessment (MoCA) <24
2. Diseases with features common to Parkinson's Disease (eg. essential tremor, multiple system atrophy, progressive supranuclear palsy)
3. Epilepsy
4. History of stroke, CVA
5. Elevated levels of ALT, AST, BUN or creatinine
6. Chronic sinusitis as defined by SNOT-20 score >1.0 on items 1-10.
7. Presence of other serious illness
8. History of brain surgery
9. History of structural brain damage
10. History of intranasal telangiectasia
11. Supplementation with glutathione and agents shown to increase glutathione will not be permitted and will require a 90 day washout period.
12. Pregnant or at risk of becoming pregnant.

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-07; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Determination of Safety | 12 weeks
  1a. Laboratory monitoring for adverse events will include CBC, ALT, AST, BUN, creatinine, uric acid, and urinalysis. Data will be collected throughout the 12-week intervention and at 1-mo following cessation of the study medication.
  1b. Clinical adverse events will be measured using a daily patient diary and record score cards specifically screening for sinus irritation. Monitoring of Side Effects System (MOSES) will be used to screen for systemic and generalized adverse events.
  1c. Effect on PD symptoms will be measured by the UPDRS to screen for accelerated disease activity.
Determination of Tolerability | 12 weeks
  Participants will be asked to keep a daily log and unused study medication will be measured at each clinical visit. Tolerability will be measured by frequency and severity of reported adverse events and withdrawal from study. The goal will be to identify the maximum tolerated dose (MTD) which will be defined as the highest dose achieving adherence, as defined as 80% of the group taking the prescribed dose 80% of the time.

SECONDARY OUTCOMES:
Description of systemic absorption characteristics | 12 weeks
  Red blood cell GSH levels will be measured at baseline, 4 weeks, and 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Mischley, ND, Principal Investigator — Bastyr University
Locations (1):
- Bastyr Clinical Research Center, Kenmore, Washington, United States